CLINICAL TRIAL: NCT01385410
Title: Effectiveness of a Baby-friendly Hospital Based Mothers' Support Group, and a Cell-phone Based Peer Support Program in Supporting Exclusive Breastfeeding in an Urban Kenyan Community.
Brief Title: Providing Peer Mother Support Through Cell Phone and Group Meetings to Increase Exclusive Breastfeeding in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Egerton University (Other); University of California, Davis (Other); Global Alliance for Improved Nutrition (Other); Emory University (Other)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 26370
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Breastfeeding
Keywords: breastfeeding exclusively
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPS, cell phone based peer support (Active Comparator): Cell phone base peer mother support for continued exclusive breastfeeding
  Interventions: Behavioral: Peer mother support for continued exclusive breastfeeding
- PSG, group meeting based peer support (Active Comparator): Group based peer Cell phone base peer mother support for continued exclusive breastfeeding
  Interventions: Behavioral: Peer mother support for continued exclusive breastfeeding
- Control (No Intervention): Current standard of care and support (national health system)

INTERVENTIONS:
Behavioral: Peer mother support for continued exclusive breastfeeding — Peer counselling on breastfeeding beginning in third trimester and continuing until 3 months postpartum
  Arms: CPS, cell phone based peer support; PSG, group meeting based peer support

SUMMARY:
This behavioural support intervention trial will investigate the potential to increase exclusive breastfeeding rates in an urban Kenyan community through peer mother support delivered either by cell phone or through group meetings. It will follow a cohort of more than 800 women attending antenatal care at a large public hospital, and compare indicators of breastfeeding and infant and maternal health between groups receiving one or other type of peer mother support. The main part of the study will test the primary hypothesis that peer group and cell phone based support can both increase rates of EBF at 3 months by 20% relative to a control group.

DETAILED DESCRIPTION:
The general objective was to assess whether participation from late pregnancy through to 3 months postpartum in bi-weekly cell phone based peer support (CPS) or monthly peer-led support groups (PSG) can increase adoption and duration of EBF amongst low-income women in Kenya served by a nationalized BFHI certified hospital above benchmarks achieved with current approaches and standard of care by existing facility-based support (SOC).

The study aimed to reach the following specific objectives related to message delivery on EBF:

assess the feasibility of two innovative approaches (CPS and PSG) to deliver extended postnatal peer support for EBF by women in an urban, low-income country setting; compare the effectiveness of these two innovative approaches to existing facility-based support; and compare the relative effectiveness of each type of peer support intervention.

ELIGIBILITY:
Inclusion Criteria for mothers:

1. attending antenatal care services at the target facility;
2. confirmed pregnant by a health care worker;
3. 24-32 weeks gestation at enrollment;
4. competency in KiSwahili or English (or both)
5. current resident of Nakuru municipality and expecting to reside there for the next 6 months;
6. intend to breastfeed their newborn;
7. self-report of any condition preventing the subject from breastfeeding (excluding HIV infection)
8. no history of mental illness
9. either HIV-negative on test result OR referred bto PMTCT services following verified positive HIV-test results
10. willing to participate in study described in IC forms
11. 18-45 years of age

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 823 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
exclusive breastfeeding | 3 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sellen, PhD, Study Director — University of Toronto; Elizabeth Kamau-Mbuthia, PhD, Principal Investigator — Egerton University; Samwel Mbugua, MSc, Principal Investigator — Egerton University; Aimee Webb Girard, Principal Investigator — Emory University
Locations (1):
- Nakuru Provincial General Hospital, Nakuru, Rift Valley, Kenya